CLINICAL TRIAL: NCT06689683
Title: Comparison of Two Different Fluoroscopy Activation Intervals in Shock Wave Lithotripsy: a Prospective Randomised Study
Brief Title: Fluoroscopy Activation Interval in SWL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lütfi Kırdar City Hospital (Other)
Responsible Party: Principal Investigator, Cengiz Canakcı, MD, Principal investigator, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Canakci0001
Record Dates: First submitted 2024-11-09; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Kidney Calculi
Keywords: kidney stone; shock wave lithotripsy; radiation
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 250 shocks (Active Comparator): In our clinic, it is standard practice to perform a fluoroscopic check after every 250 shocks during the SWL session. Group 1 was fluoroscopically monitored every 250 shocks.
  Interventions: Device: Shock wave lithotripsy
- 500 shocks (Active Comparator): Group 2 was fluoroscopically monitored every 500 shocks.
  Interventions: Device: Shock wave lithotripsy

INTERVENTIONS:
Device: Shock wave lithotripsy — SWL works on the principle of focusing on the calculus using fluoroscopy. There has yet to be a consensus on the optimal frequency of fluoroscopic monitoring in the literature.

SUMMARY:
Shock wave lithotripsy (SWL) is a noninvasive method widely used as the first step in treating stone disease. This study aimed to reduce radiation exposure to patients and practitioners during SWL sessions by extending the intervals of fluoroscopy controls. The main questions it aims to answer are:

* Will radiation exposure be reduced?
* Will the stone-free status be affected? The researchers will compare the fluoroscopic control intervals of 250 shocks and 500 shocks.

Participants will:

* Take to a maximum of 3 sessions.
* Check once a week
* Group 1 was fluoroscopically monitored every 250 shocks, and Group 2 was fluoroscopically monitored every 500 shocks

DETAILED DESCRIPTION:
SWL works on the principle of focusing on the calculus using ultrasonography or fluoroscopy, transmitting high-energy shock waves from the lithotripter to the calculus and fragmenting it. Fluoroscopic focusing is a commonly used imaging technique that raises concerns about ionizing radiation exposure for patients, technologists, and physicians. Intermittent fluoroscopic monitoring during SWL is widely employed to adjust for patient movement, respiratory movement, and stone displacement within the kidney. However, there is no consensus on the optimal frequency of fluoroscopic monitoring in the literature. This study aims to seek to determine whether increasing the duration between fluoroscopic checks affects the success rate of SWL in achieving stone-free status while reducing radiation exposure to patients.

ELIGIBILITY:
Inclusion Criteria:

* radiopaque renal pelvic stones smaller than 2 centimeters.

Exclusion Criteria:

* anatomical anomalies, coagulation disorders, non-opaque calculi, active urinary infection and distal obstruction

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2020-07-27 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
evaluate The effect of two different fluoroscopic activation intervals on the stone-free rate. | 1 month after the end of treatment
  Session intervals were determined as one week, and patients with residues visible on the KUB radiography before the session were included in the new session. At the end of the treatment, direct radiography and ultrasound of the urinary system was performed at the end of the first month. Patients with stones larger than 4 mm were considered to have had an unsuccessful treatment.

SECONDARY OUTCOMES:
Secondary endpoints were total fluoroscopy time and complications. | From registration until the 1st month after the end of treatment.
  The total fluoroscopy time (seconds) during treatment will be calculated.
Secondary endpoints were complications. | From registration until the 1st month after the end of treatment.
  Complications occurring from the beginning of treatment to the end of treatment, such as additional intervention, pyelonephritis, steinstrausse.

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University Kartal Dr. Lütfi Kırdar City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No